CLINICAL TRIAL: NCT01154309
Title: Group Cognitive Behavioral Therapy for Depression and Alcohol and Other Drug Disorders
Brief Title: Group CBT for Depression and AOD Disorders
Acronym: BRIGHT2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Behavioral Health Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01DA020159 (NIH)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Depression; Substance Use
Keywords: Depression; Substance Use; Group Cognitive Behavioral Therapy
MeSH Terms: conditions — Depression; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Clients are invited to attend 18 group CBT sessions
  Interventions: Behavioral: Group CBT for Depression and AOD Disorders
- 2 (No Intervention): Clients receive usual care

INTERVENTIONS:
Behavioral: Group CBT for Depression and AOD Disorders — 18 sessions of 2-hour group CBT
  Arms: 1

SUMMARY:
The investigators will adapt and test an existing treatment (group CBT for depression) for use in outpatient substance use treatment settings as delivered by trained substance use counselors. The investigators expect that treatment will lead to improved depression and substance use outcomes.

DETAILED DESCRIPTION:
Aim 1. To adapt an existing group therapy (CBT for depression), creating a manualized treatment and accompanying implementation measures and tools for use with clients with persistent depressive symptoms and AOD disorders and to obtain preliminary assessments of the treatment from patient and provider perspectives.

Aim 2. To conduct a pilot test of the revised treatment in which we (a) demonstrate that when the therapy is implemented with fidelity, clinically significant reductions in depressive symptoms and AOD use occur; (b) estimate the likely effect size; and (c) investigate the underlying mechanisms of change, including both cognitive-behavioral and group processes and their relationship to depression and AOD treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in outpatient substance abuse program
* BDI II score >13
* Probable alcohol or substance use problem

Exclusion Criteria:

* Cognitive impairment (Short Blessed > 10)
* Probably bipolar or schizophrenic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Reductions in depressive symptoms as measured by the BDI II | Post treatment
Reductions in AOD use | Post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Watkins, MD, MSHS, Principal Investigator — RAND
Locations (1):
- Behavioral Health Services, Inc, Gardena, California, United States